CLINICAL TRIAL: NCT05286177
Title: Does Volume-based Enteral Feeding Improve Nutrient Delivery in Hospitalized Critically Ill Children? a Randomized Feasibility Trial of Volume Versus Rate-based Enteral Nutrition Algorithms.
Brief Title: Does Volume-based Enteral Feeding Improve Nutrient Delivery in Hospitalized Critically Ill Children?
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: American Society for Parenteral and Enteral Nutrition (Other); Alberta Health services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REB21-0773
Record Dates: First submitted 2022-01-04; First posted 2022-03-18 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Enteral Feeding

STUDY DESIGN:
Intervention Model Description: The investigators will conduct a single-center parallel partially blinded 1:1 randomized feasibility trial of 20 children admitted to the Alberta Children's Hospital (ACH) PICU.
Who Masked: Investigator, Outcomes Assessor
Masking Description: A double-blinded strategy is not feasible for this study because the medical team cannot remain adequately blinded to study arms after randomization. Bedside nurses delivering EN support need to know which feeding algorithm to follow. The medical team (including PICU physicians, nurse practitioners, and dietitians) have access to patients' medical records which include current hourly infusion rates of enteral feeds so they will be able to deduce the patients' allocations. The team uses current hourly infusion rates to assess fluid balance and to make clinical decisions.
  To minimize bias, the research assistant tasked with data collection will remain blinded to study allocation throughout data collection and will enter the data into the REDCap Database in a blinded fashion. After data collection and prior to data analysis, all identifying information will be saved in a separate file to ensure the Study Coordinator will be re-blinded to participant allocation during data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Volume-based EN (Experimental): Volume-based EN algorithm arm.
  Interventions: Procedure: Volume-based EN
- Rate-based EN (Active Comparator): Rate-based EN algorithm (standard of care).
  Interventions: Procedure: Rate-based EN

INTERVENTIONS:
Procedure: Volume-based EN — Bedside nurses will receive a total daily feed volume prescription to be administered to the participant over a 24-hour period. The bedside nurse will calculate the initial hourly rate by dividing the total daily feed goal by 24 hours at approximately 0700 hours. In this intervention group, they will be instructed to titrate the rate of feeds to accommodate for any feeding interruptions as follows: When feeds are held for > 1 hour, the remaining daily feed volume will be divided by the remaining number of hours. A maximum infusion rate will be set at 2 times the patient's baseline 24-hour feed rate to ensure that a large bolus volume of feed is not administered over a too short period of time.
  Arms: Volume-based EN
Procedure: Rate-based EN — Bedside nurses will receive an hourly feed rate prescription to administer the tube feedings over a 24-hour period. If feeds are held, they will be restarted at the same consistent hourly rate that was previously ordered. Nurses will not adjust feed rates to compensate for feed interruptions
  Arms: Rate-based EN

SUMMARY:
Background Some critically ill children have malnutrition which may worsen while they are in hospital and delay their return home. They can recover faster when they are given tube feedings to improve their nutrition. Unfortunately, in the hospital these feedings are often interrupted and so these children do not get all the nutrition they need. The usual procedure is to set hourly rates for the tube feedings and to accept that they get less when feedings are interrupted. The researchers would like to test if children are fed better if the bedside nurses were to check the volume provided through the day and then ensure the child gets closer to the prescribed volumes.

Aim To determine the feasibility of performing a Randomized Control Trial assessing the use of a Volume-based feeding algorithm in critically ill children admitted to the Alberta Children's Hospital Pediatric Intensive Care Unit (PICU).

Objectives

1. Obtain information to inform sample size calculations for nutrition and clinical outcomes for a larger RCT: energy adequacy and protein adequacy, feed tolerance, infections, changes in anthropometric measurements at transitions of care, 28-day ventilator free days, length of stay, 60-day mortality, and 60-day hospital readmission?
2. Assess adherence of medical staff to the study protocol
3. Evaluate the timing of study enrollment and participant allocation
4. Evaluate the proposed deferred consent strategy.

Methods The researchers will conduct a randomized control feasibility trial of critically ill children admitted to the Alberta Children's Hospital (ACH) Pediatric Intensive Care unit who require tube feedings. Children will be randomly assigned to the intervention arm (Volume-based algorithm) or the comparison arm (rate-based algorithm).

Significance The proposed study will provide evidence of whether a novel approach to feeding critically ill children is feasible during PICU admission. This trial will inform a larger Randomized Control Trial on this topic that will assess if using a Volume-based feeding algorithm will improve outcomes of clinical importance including energy adequacy, protein adequacy, feed tolerance, infections, changes in anthropometric measurements at transitions of care, 28-day ventilator free days, length of stay in PICU and hospital, 60-day mortality, and 60-day hospital readmission.

DETAILED DESCRIPTION:
Malnutrition is prevalent in hospitalized critically ill children, may worsen throughout hospital admission, and is associated with negative outcomes including increased ventilator days and longer hospital stays. Early optimal enteral nutrition (EN) is associated with improved outcomes including reduced mortality and shorter hospital stays. Unfortunately, feed interruptions are common which result in underfeeding and accumulating nutrient deficits. Traditionally in pediatrics, tube feedings are ordered and provided using hourly rate-based EN algorithms, which direct the nurse to run the feeding pump at a prescribed hourly rate. The problem with this approach is that the nurse is not authorized to compensate for feed interruptions. Using a daily volume-based EN goal would circumvent this issue by allowing bedside nurses to adjust feedings to be able to deliver the 24-hour desired goal and compensate for feed disruptions. Research conducted in adult critical care comparing volume based versus rate based EN algorithms have shown superior energy and protein delivery. To the researchers knowledge, no pediatric studies have compared volume to rate-based EN.

Aim To determine the feasibility of performing a randomized controlled trial (RCT) assessing the use of a volume-based versus rate-based feeding algorithm in critically ill children admitted to the pediatric intensive care unit (PICU).

Objectives

The primary objective is to assess the feasibility of the proposed randomized control trial to evaluate a Volume-based EN algorithm in the PICU by:

Assessing participant enrollment and recruitment Assessing adherence of medical and nursing staff to the study protocol Evaluating the acceptability of the proposed deferred consent strategy The secondary objective will be to obtain data to inform sample size calculations for nutrition (energy and protein adequacy) and clinical outcomes (feed tolerance, infections, changes in anthropometric measurements at transitions of care, 28-day ventilator free days, length of stay, 60-day mortality, and 60-day hospital readmission) for the larger RCT.

Methods: The investigaters will conduct a single-center parallel partially-blinded 1:1 randomized feasibility trial of 20 children admitted to the Alberta Children's Hospital PICU. Children/adolescents aged 1 month to 18 years, who the investigators anticipate will be admitted to the PICU for ≥ 48 hours, and who initiate enteral nutrition support will be eligible. The trial will compare a volume-based EN algorithm (intervention) to the standard of care rate-based EN algorithm (control). Randomization will be block-stratified by age and ventilator status (invasive ventilation or other). The clinical team will remain unblinded to group allocation to be able to perform care. The research team will remain blinded to allocation to minimize bias.

Adherence to study protocol will be assessed as the number of times that medical or nursing staff deviate from the allocated feeding algorithm.

Enrollment and recruitment of participants will be evaluated by assessing the proportion of eligible participants who are successfully enrolled into the study. Reasons for non-enrollment will be recorded.

Deferred Consent: There is growing evidence that requesting consent close to admission into a PICU puts undo stress on parents/caregivers which can result in limited study enrollment. Deferred consent allows us to randomize eligible children at the time of the decision to use tube feedings and to start the study intervention prior to obtaining consent. This approach provides time to approach caregivers when they are not dealing with the fact that their child has been admitted to intensive care. As far as the investigators are aware, there is no evidence for using a deferred consent model in an enteral feeding RCT. Therefore, part of this feasibility study will assess this strategy for nutrition care research. Quantitative evaluation will be used to estimate the length of time it takes between randomization of eligible participants to starting the assigned feeding algorithm to obtaining consent/assent, the proportion of eligible subjects who provide consent/assent, and any concerns raised. Qualitative methods using the Theoretical Domains Framework will be used to assess parents' perceptions and experiences related to the deferred consent strategy using semi-structured interviews.

Baseline data collected will include age, sex, PRISM IV score (severity of illness), admission diagnosis, and admission comorbidities. Anthropometrics will be measured as soon as possible after PICU admission and at transfer to another unit and/or to home. Data for sample size estimations will be collected prospectively including daily prescribed calories and protein, daily received calories and protein, feed intolerance, deviations from assigned algorithm, ventilator days, days with inotropic support, and length of stay and mortality at PICU and hospital discharge will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Children 1-month post-natal age to 18 years of age
* Children anticipated by the intensivist or nurse practitioner to be admitted to the PICU for ≥ 48 hours
* Children who will be initiated on EN support

Exclusion Criteria:

* Children will not be eligible for this study if they are palliative
* Children who have contraindications to EN (i.e., a non-functional GI tract)
* Children who are on parenteral nutrition
* Children who are being fed by a bolus feed regime
* Children who cannot progress past trophic feed volumes within 24 hours of EN initiation
* Children anticipated to be admitted to PICU for <48 hours

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Assess participant enrollment and recruitment will be completed by documenting the number of children who successfully initiate the study protocol. | Up to 12 months
  The investigators will evaluate the proposed inclusion/exclusion criteria, participant recruitment, and enrollment. On weekdays, during bedside rounds, the study coordinator will assess eligibility of admitted children against the inclusion/exclusion criteria. On Mondays the Study Coordinator will compare patients who were admitted over the weekend with the inclusion/exclusion criteria. After randomization, the number of children The investigators will evaluate the proposed inclusion/exclusion criteria, participant recruitment, and enrollment.
Number of deviations from assigned feeding algorithm. | Up to 12 months
  The Research Assistant will document if a deviation from the allocated feeding algorithm (volume-based or rate-based) occurred in the study database daily while participants are being fed via the research protocol.
Reason for participant attrition/withdraw from study. | Up to 12 months
  The research assistant will document the reason for participant removal from the study protocol in the secure REDcap database.
Day of participant attrition/withdraw from study. | Up to 12 months
  The research assistant will document the study day of participant removal from the study protocol in the secure REDcap database.
The length of time it takes between randomization of eligible participants to starting the assigned feeding algorithm to obtaining consent/assent. | Up to 12 months
  The time that randomization of an eligible participant occurs and the time that the participant starts the assigned feeding alogirhtm and the time that the Research Coordinator obtains consent/assent will be recorded.
Proportion of eligible subjects who provide consent/assent. | Up to 12 months
  The number of eligible subjects who provided consent/assent and the number who declined consent/assent will be recorded and used to assess the proportion of subjects who provide consent.
10 semi structured qualitative interviews to to assess guardians/caregiver perception and experiences around deferred consent. | Semi-structured interviews will take place after PICU discharge - up to 6 months
  Participants will be selected through purposive sampling of parents/guardians of patients enrolled in both arms of the EN trial. Zoom semi-structured interviews will be conducted. Interviews will be recorded for data analysis. A minimum sample size for interviews set a-priori will be 10, with additional interviews theme saturation in reached. Data collection will be stopped once no new themes emerge.
10 semi structured qualitative interviews to to assess patient experiences around deferred consent. | Semi-structured interviews will take place after PICU discharge - up to 6 months
  Participants will be selected through purposive sampling of patients enrolled in both arms of the EN trial. Zoom semi-structured interviews will be conducted. Interviews will be recorded for data analysis. A minimum sample size for interviews set a-priori will be 10, with additional interviews theme saturation in reached. Data collection will be stopped once no new themes emerge.

SECONDARY OUTCOMES:
Calories received - (daily total kcal) | Up to 12 months
  This will be used to calculate energy adequacy by dividing daily total calories recieved by prescribed energy goal based on WHO BMR equations or indirect calorimetry.
Protein received - (daily total grams protein) | Up to 12 months
  This will be used to calculate protein adequacy by dividing daily total grams protein received by goal prescribed protein based on CCSM/ASPEN guidelines.
Enteral feeding route use - gastric or post-pyloric | Up to 12 months
  Research assistant will find this information in the electronic medical record.
Participant height in centimeters | Within 48 hours of PICU admission, within 48 hours of PICU discharge and within 48 hours of hospital discharge.
  Height in cm will be measured at three time points - admission to PICU, discharge from PICU and discharge from hospital
Participant weight in kilograms | Within 48 hours of PICU admission, within 48 hours of PICU discharge and within 48 hours of hospital discharge.
  Weight in kg will be measured at three time points - admission to PICU, discharge from PICU and discharge from hospital
Mid upper arm circumference in cm in children >6 months of age | Within 48 hours of PICU admission, within 48 hours of PICU discharge and within 48 hours of hospital discharge.
  MUAC will be measured at three time points - admission to PICU, discharge from PICU and discharge from hospital
Number of days of PICU admission when feed intolerance occurs will be recorded. | Daily throughout PICU admission up to 12 months
  Feed intolerance in a 24-hour period will be defined as new onset >2 episodes of diarrhea, >2 episodes of emesis, and/or abdominal distention that results in holding feeds.
Number of days on invasive ventilation | Daily throughout PICU admission up to 12 months
  Days when a participant is being invasively ventilated will be recorded by the research assistant.
Number of days in PICU on non-invasive ventilation | Up to 12 months while in PICU
  Days when a participant is on non-invasive ventilatory support will be recorded by the research assistant.
Number of days in PICU on nasal prongs (high flow O2 or low flow O2) | Up to 12 months while in PICU
  Days when a participant is on high flow O2 or low flow O2 will be recorded by the research assistant.
Number of days in PICU on inotrope medications | Up to 12 months while in PICU
  Vasoacctive medications including but not limited to epi, norepi, dopamine
Number of episodes of culture positive infections | Up to 12 months while in PICU
  Each culture positive infection (blood stream, speutum) will be documented as a separate event.
PICU length of stay (days) | Up to 12 months while in PICU
  Number of days a participant is admitted to PICU will be recorded by the research assistant.
Hospital length of stay (days) | Up to 12 months while admitted to any unit at ACH
  Number of days a participant is admitted to the Alberta Children's Hospital will be recorded by the research assistant.
Ventilator free days | Up to 12 months while in PICU
  The number of ventilator free days, defined as days alive and free from invasive ventilation, will be collected from PICU admission to 28 days after admission.
PICU mortality | Up to 12 months while in PICU
  If a participant dies while admitted to ACH PICU this will be recorded.
Hospital mortality | Up to 12 months while in admitted to ACH
  During current admission
60-day PICU mortality | Up to 60 days from admission to PICU
  If a participant dies up to 60 days after PICU admission day 1.
60-day readmission to hospital | Up to 60 days from admission to PICU
  If a participant is readmitted within 60 days of discharge from ACH.
Pediatric Risk of Mortality score (PRISM IV) | Up to 12 months
  PRISM IV score is a severity of illness score which is calculated at admission to PICU. PRISM IV provides a prediction of mortality and as the score increases chance of mortality increases.
Admission diagnosis | Up to 12 months
  reason for admission to PICU
Admission Comorbidities | Up to 12 months
  Comorbidities present at time of admission to PICU

CONTACTS AND LOCATIONS:
Overall Officials: Tanis Fenton, PhD, Principal Investigator — University of Calgary
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No